CLINICAL TRIAL: NCT02510092
Title: In Vivo Intravascular Diagnostics and Evaluation of New Therapeutic Modalities in Systemic Autoimmune and Coronary Artery Disease Patients
Brief Title: Coronary Artery and Systemic Autoimmune Disease: Diagnostics and Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Semmelweis University Heart and Vascular Center (Other)
Collaborators: University of Debrecen (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Im-CAD-001
Record Dates: First submitted 2015-07-23; First posted 2015-07-28 (Estimated); Last update posted 2021-04-23 (Actual); Status verified 2021-04

CONDITIONS: Autoimmune Diseases; Coronary Artery Disease
MeSH Terms: conditions — Autoimmune Diseases; Coronary Artery Disease | interventions — Percutaneous Coronary Intervention

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Coronary artery diseae with revascularization indicated (Active Comparator): Subjects with coronary artery disease, that require and are eligible for percutaneous revascularization.
  Interventions: Device: Percutaneous coronary intervention with new generation fully resorbable scaffold
- Coronary artery disease not requiring revascularization (No Intervention): Subjects with coronary artery disease that do not require revascularization.

INTERVENTIONS:
Device: Percutaneous coronary intervention with new generation fully resorbable scaffold
  Arms: Coronary artery diseae with revascularization indicated

SUMMARY:
This study evaluates in vivo intracoronary imaging using intravascular ultrasound and optical coherence tomography and safety and efficacy of new generation fully bioresorbable vascular scaffolds in four well defined systemic autoimmune (rheumatoid arthritis, mixed connective tissue disease, systemic sclerosis, systemic lupus erythematosus) and concomitant coronary disease patients.

DETAILED DESCRIPTION:
The aim of this study is to assess in vivo intracoronary anatomy using intravascular ultrasound and optical coherence tomography and assess the efficacy and safety of new generation fully bioresorbable vascular scaffolds in a systemic autoimmune and coronary heart disease patient population.

The following four well defined systemic autoimmune entities are linked to increased cardiovascular risk: rheumatoid arthritis, mixed connective tissue disease, systemic sclerosis and systemic lupus erythematosus. One of the main causes of death in systemic autoimmune subjects is cardiovascular disease. In-vivo intracoronary anatomy and pathology regarding systemic autoimmune diseases is unknown. Furthermore, all forms of revascularization in such patients yield sub-optimal results, with poor outcomes using even the most modern drug eluting metallic stents. This may be linked to a long term exaggerated chronic inflammation response to the metallic components. Thus, fully bioresorbable vascular scaffolds may prove more efficacious in systemic autoimmune subjects.

ELIGIBILITY:
Inclusion Criteria:

* Age of 18+ years
* Signed and dated informed consent form
* Manifest autoimmune disease, consisting either of: rheumatoid arthritis or systemic lupus erythematosus or systemic sclerosis or mixed connective tissue disease under the care of a clinical immunologist
* Clinical indication for a coronary angiography as determined by a cardiologist

Exclusion Criteria:

* Age of 75+ years
* Glomerular filtration rate of under 30 ml/min
* Severely decreased left ventricular function (ejection fraction <35%)
* Pregnancy or nursing
* Unclear immunological diagnosis

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2015-07; Primary Completion 2021-03 (Actual); Study Completion 2021-03 (Actual)

PRIMARY OUTCOMES:
Major adverse cardiac and cerebral events | From index procedure to 5 years
  Eligible for patients in clinical need for revascularization undergoing percutaneous revascularization with a bioresorbable vascular scaffold

OTHER OUTCOMES:
Intravascular ultrasound findings in coronaries | At index procedure
  Minimum Lumen Area (MLA)
Intravascular ultrasound findings in coronaries | At index procedure
  Percent Atheroma Volume (PAV)
Intravascular ultrasound findings in coronaries | At index procedure
  Area Stenosis (AS)
Intravascular ultrasound findings in coronaries | At index procedure
  Negative or positive remodelling index (RI)
Intravascular ultrasound findings in coronaries | At index procedure
  Intimal thickness (IT)
Intravascular ultrasound findings in coronaries | At index procedure
  Calcification Index (CI)
Optical coherence tomography findings in coronaries | At index procedure
  Intima to Media ratio (I/M ratio)
Optical coherence tomography findings in coronaries | At index procedure
  Excentric intima hyperplasia
Optical coherence tomography findings in coronaries | At index procedure
  Thin Cap Fibroatheroma presence (TCFA)
Optical coherence tomography findings in coronaries | At index procedure
  Macrophage infiltration
Optical coherence tomography findings in coronaries | At index procedure
  Intramural hematoma formation
Optical coherence tomography findings in coronaries | At index procedure
  Intimal laceration
Optical coherence tomography findings in coronaries | At index procedure
  Microchannel formation
Optical coherence tomography findings in coronaries | At index procedure
  Lipid pool formation

CONTACTS AND LOCATIONS:
Locations (1):
- Semmelweis University Heart and Vascular Center, Budapest, Hungary